CLINICAL TRIAL: NCT01032382
Title: Double-blind, Randomized, Pharmacokinetics, Safety, and Efficacy Trial of WR 279,396 (Paromomycin + Gentamicin Topical Cream) and Paromomycin Topical Cream for the Treatment of Cutaneous Leishmaniasis in Peru
Brief Title: Safety, Efficacy and Pharmacokinetics (PK) Study of WR 279,396 Versus Paromomycin for Treatment of Cutaneous Leishmaniasis (Peru-PK)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PG-PERU-08-03, A-15809
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2014-08

CONDITIONS: Leishmaniasis, Cutaneous
Keywords: leishmaniasis; cutaneous; WR 279,396; paromomycin; gentamicin; pharmacokinetics; safety; efficacy
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Leishmaniasis | interventions — Paromomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paromomycin Alone Treatment (Active Comparator)
  Interventions: Drug: Paromomycin Alone Cream (15% paromomycin topical cream)
- WR 279,396 (Active Comparator)
  Interventions: Drug: WR 279,396 (15% paromomycin + 0.5% gentamicin topical cream)

INTERVENTIONS:
Drug: WR 279,396 (15% paromomycin + 0.5% gentamicin topical cream) — topical application to CL lesions once daily for 20 days
  Other Names: Topical paromomycin/gentimicin cream
  Arms: WR 279,396
Drug: Paromomycin Alone Cream (15% paromomycin topical cream) — topical application to CL lesions once daily for 20 days
  Arms: Paromomycin Alone Treatment

SUMMARY:
The objectives of the study are to evaluate the pharmacokinetics (PK), safety, and efficacy of WR 279,396 (Paromomycin + Gentamicin Topical Cream) and Paromomycin Topical Cream in subjects with cutaneous leishmaniasis (CL).

DETAILED DESCRIPTION:
This study is a single-site, randomized, double-blind, two group trial assessing the PK, safety and efficacy of WR 279,396 Topical Cream and Paromomycin Topical Cream in subjects with CL. Subjects will be screened over a period up to 28 days for eligibility including parasitology for confirmation of ulcerative CL. Subjects will be randomized in a targeted 1:1 ratio to receive either WR 279,396 (15% paromomycin + 0.5% gentamicin topical cream) (target n=15) or Paromomycin Topical Cream (15% paromomycin topical cream) (target n=15) by topical application to CL lesions once daily for 20 days. Because the primary objective of this trial is to determine PK in all age groups, subjects will be stratified by age: 5-11 yrs, 12-17 yrs, and ≥ 18 yrs with at least 6 PK subjects in each age stratum and no more than 18 total subjects will be randomized in any age range. A target of 30 subjects who complete the PK part of the study is the goal. Any subject who does not complete the PK portion of the study will be replaced with another subject from the same age group that will be given the same treatment assignment to maintain the balance. Safety will be assessed by monitoring adverse events (AEs), lesion site reactions, vital signs, and blood creatinine levels. The primary efficacy analysis will be by evaluation of an index lesion with secondary efficacy analyses including all lesions. Lesions will also be examined for parasite negativity by classical means (positive culture for promastigotes or microscopic identification of amastigotes in stained lesion tissue) on Day 21.

In adult subjects, on Days 1 and 20, blood will be collected prior to topical cream application and at 0.5h, 1h, 2h, 3h, and 4h ± 5 minutes and 8h, 12h, and 24h ± 15 minutes after completion of cream application to determine plasma levels of paromomycin and gentamicin to calculate PK parameters. Thus, the last blood draw in this series will occur on Day 21. In addition, blood will be collected on Days 4, 7, 12, and 17 ± 1 day before study drug application to examine trough plasma levels of paromomycin and gentamicin. A follow-up plasma sample for PK analysis will also be obtained on Day 28 ± 2 days.

Subjects under the age of 18 years will have a total of four blood samples drawn. The first will be drawn at pre-application and the second will be drawn at 4 hours ± 5 minutes after completion of application of the topical cream on Study Day 1. The third will be drawn pre-application and the fourth at 4 hours ± 5 minutes after completion of application of the topical cream on Study Day 20. Subjects who receive Paromomycin Topical Cream are not expected to have blood levels of gentamicin, but as the study is blinded, plasma specimens will be tested for both paromomycin and gentamicin.

The index lesion (primary ulcerated) and all other ulcerated lesions will be assessed for clinical response by measurement of the length and width of area of ulceration. A lesion will be considered to be completely cured if 100% re-epithelialization is observed (i.e., this is a measurement of ulceration of 0 x 0 mm). Non-ulcerated lesions will also be measured to monitor the total area of exposure of lesions to study drug and will be evaluated for cure (i.e., absence of signs of an active lesion).

Subjects will have an in-clinic follow-up weekly (Days 28, 35, 42, 49, 56, and 63 ± 2 days) after completion of treatment for safety assessments, lesion measurements, and lesion photographs. On Day 21, index lesions in adult subjects that have not completely re-epithelialized will be assessed for parasites by classical means (positive culture for promastigotes or microscopic identification of amastigotes in stained lesion tissue). An interim analysis of all of the data collected on all subjects who were randomized and completed the nominal Day 63 follow-up will be performed to make decisions about the final design of a Phase 3 trial. Subjects will continue to be followed for outcomes at Day 100 and 168 ± 14 days. A final analysis of outcomes after the longer term followup period has been completed for all subjects will be performed when the trial is closed. Follow-up evaluations include AEs, medication use, lesion measurements, and lesion photographs.

Patients who fail therapy (see definition of failure below) may be administered rescue therapy at the discretion of the patient's personal physician.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the study, the following must be answered "YES" or not applicable, as appropriate for the study subject:

  1. Is the subject a male or female at least 5 years-of-age?
  2. Is the subject or legal guardian able to give written informed consent or assent, as appropriate?
  3. Does the subject have a diagnosis of CL in at least one lesion by at least one of the following methods: 1) positive culture for promastigotes, or 2) microscopic identification of amastigotes in stained lesion tissue.
  4. Does the subject have at least one ulcerative lesion ≥ 1 cm and ≤ 5 cm, that meets the criteria for an index lesion?
  5. Is the subject willing to forego other forms of treatments for CL including other investigational treatments during the study?
  6. In the opinion of the investigator, is the subject (or their legal guardian) capable of understanding and complying with the protocol?
  7. If female and of child-bearing potential, did the subject have a negative pregnancy test during screening and agree to use an acceptable method of birth control during the treatment phase and for 1 month after treatment is completed?
  8. Does the subject have adequate venous access for blood draws?

Exclusion Criteria:

To be eligible for the study, the following must be answered "NO" or not applicable as appropriate for the study subject:

1. Does the subject have only a single lesion whose characteristics include any of the following: verrucous or nodular lesion (non-ulcerative), lesion <1 cm in its greatest diameter, lesion in a location that in the opinion of the Investigator is difficult to maintain application of study drugs topically?
2. Does the subject have a lesion due to leishmania that involves the mucosa or palate or any signs of mucosal disease that might be due to leishmania?
3. Does the subject have signs and symptoms of disseminated disease in the opinion of the Principal Investigator?
4. Does the subject have > 10 lesions?
5. Is the subject a female who is breast-feeding?
6. Does the subject have an active malignancy or history of solid, metastatic or hematologic malignancy with the exception of basal or squamous cell carcinoma of the skin that has been removed?
7. Does the subject have significant organ abnormality, chronic disease such as diabetes, severe hearing loss, evidence of renal or hepatic dysfunction, or creatinine greater than 15%, or aspartate aminotransferase (AST), or alanine aminotransferase (ALT) greater than 1.5 times the above the upper limit of normal (ULN) as defined by the clinical laboratory defined normal ranges?
8. Has the subject received treatment for leishmaniasis including any medication with pentavalent antimony including sodium stibogluconate (Pentostam), meglumine antimoniate (Glucantime); amphotericin B (including liposomal amphotericin B and amphotericin B deoxycholate); or other medications containing paromomycin (administered parenterally or topically) or methylbenzethonium chloride (MBCL); gentamicin; fluconazole; ketoconazole; pentamidine; miltefosine, azithromycin or allopurinol that was completed within 8 weeks of starting study treatments?
9. Does the subject have a history of known or suspected hypersensitivity or idiosyncratic reactions to aminoglycosides?
10. Does the subject have any other topical disease/condition which would interfere with the objectives of this study?

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Llanos-Cuentas, M.D., Principal Investigator — Universidad Peruana Cayetano Heredia (UPCH)
Locations (1):
- Universidad Peruana Cayetano Heredia (UPCH), Lima, Peru

REFERENCES:
- [Derived] Ravis WR, Llanos-Cuentas A, Sosa N, Kreishman-Deitrick M, Kopydlowski KM, Nielsen C, Smith KS, Smith PL, Ransom JH, Lin YJ, Grogl M. Pharmacokinetics and absorption of paromomycin and gentamicin from topical creams used to treat cutaneous leishmaniasis. Antimicrob Agents Chemother. 2013 Oct;57(10):4809-15. doi: 10.1128/AAC.00628-13. Epub 2013 Jul 22. PMID 23877689

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Started | 16 | 14
Completed | 11 | 9
Not Completed | 5 | 5
Not completed — Disease dissemination | 1 | 1
Not completed — Treatment failure | 3 | 1
Not completed — Index lesion relapse | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paromomycin Alone Treatment | WR 279,396 | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.7 (16.2) | 18.2 (15.1) | 19.5 (15.5)
Age, Customized [Number; unit: participants]
  Adults (18+ years) | 5 | 4 | 9
  Children (12 to 17 years) | 5 | 3 | 8
  Children (5 to 11 years) | 6 | 7 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Final Clinical Cure for Index Lesions
Description: Final clinical cure was defined as follows:
  1. Subject has initial clinical cure (100% re-epithelialization of index lesion by nominal Day 63); OR,
  2. Subject has initial clinical improvement (> 50% re-epithelialization of index lesion by nominal Day 63 followed by 100% re-epithelialization of the index lesion on or before nominal Day 100; AND,
  3. Subject has no relapse of index lesion by Day 168. Relapse was defined as an index lesion meeting the criteria for initial clinical cure that had any new ulceration/nodule (> 0 x 0 mm measurement) by nominal day 168, or an index lesion meeting the criteria for initial clinical improvement that subsequently enlarged by nominal Day 168.
Time Frame: Initial clinical cure by day 63 and no relapse by day 168
Measure: Number; unit: participants
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Number analyzed (Participants) | 16 | 14
participants | 11 | 9

2. Secondary Outcome: Detectable Paromomycin Plasma Levels
Description: Paromomycin plasma concentrations following administration of paromomycin alone or WR 279,396 in adults
Time Frame: Day 4, 7, 12, 17, 20, 28
Population: Adults (18+ years)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Number analyzed (Participants) | 5 | 4
ng/mL
  Day 4 | 12.1 (27.0) | 37.3 (74.5)
  Day 7 | 10.3 (23.1) | 17.9 (35.8)
  Day 12 | 36.2 (33.2) | 78.9 (81.6)
  Day 17 | 210.0 (327.0) | 162.0 (123.0)
  Day 20 | 87.3 (109.0) | 128.0 (58.7)
  Day 28 | 0 (0) | 0 (0)

3. Secondary Outcome: Paromomycin Plasma Concentrations in Children
Description: Paromomycin plasma concentrations 4 hours following administration of paromomycin alone or WR 279,396 in children
Time Frame: 0 and 4 hours on days 1 and 20
Population: Children ages 5 to 17 (inclusive)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Number analyzed (Participants) | 11 | 10
ng/mL
  Day 1 hour 0 | 6.2 (20.5) | 22.1 (69.9)
  Day 1 hour 4 | 71.2 (88.0) | 322.0 (757.0)
  Day 20 hour 0 | 93.8 (59.9) | 89.2 (132.0)
  Day 20 hour 4 | 744.0 (503.0) | 1030.0 (1460.0)

4. Secondary Outcome: Pharmacokinetic Parameter: Cmax
Description: Cmax of paromomycin following administration of paromomycin alone or WR 279,396 to adults in Panama
Time Frame: 0, 0.5, 1.0, 2.0, 3.0, 4.0, 8.0, 12.0, 24.0 hours on both Days 1 and 20
Population: Adults (18+ years)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Number analyzed (Participants) | 5 | 4
ng/mL
  Day 1 | 511 (445) | 155.0 (139.0)
  Day 20 | 1400 (842) | 882 (124)

5. Secondary Outcome: Pharmacokinetic Parameter: Tmax
Description: Pharmacokinetic Parameter: Tmax
Time Frame: 0, 0.5, 1.0, 2.0, 3.0, 4.0, 8.0, 12.0, 24.0 hours on both Days 1 and 20
Population: Adults (18+ years). On day 1, Paromomycin Alone Treatment group N = 4; WR 279,396 group N = 3.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Number analyzed (Participants) | 5 | 4
hr
  Day 1 | 2.25 (0.5) | 3 (1.73)
  Day 20 | 4.6 (3.13) | 3 (1.15)

6. Secondary Outcome: Pharmacokinetic Parameter: Area Under the Curve (AUC)
Description: Area under the curve (AUC) of paromomycin following administration of paromomycin alone or WR 279,396 to adults in Panama
Time Frame: 0, 0.5, 1.0, 2.0, 3.0, 4.0, 8.0, 12.0, 24.0 hours on both Days 1 and 20
Population: Adults (18+ years)
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Number analyzed (Participants) | 5 | 4
ng*hr/mL
  Day 1 | 3154 (3562) | 1228 (1413)
  Day 20 | 13331 (9156) | 8955 (1955)

7. Secondary Outcome: Pharmacokinetic Parameter: t(1/2)
Description: t(1/2) of paromomycin following administration of paromomycin alone or WR 279,396 to adults in Panama
Time Frame: 0, 0.5, 1.0, 2.0, 3.0, 4.0, 8.0, 12.0, 24.0 hours on both Days 1 and 20
Population: Adults (18+ years). WR 279,396 group measurements Day 1 N = 2 and Day 20 N = 4. One study participant in the Paromomycin Alone Treatment was withdrawn at Day 100.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Number analyzed (Participants) | 4 | 4
hr
  Day 1 | 2.55 (1.23) | 4.51 (0.06)
  Day 20 | 7.17 (3.29) | 6.81 (3.2)

8. Secondary Outcome: Pharmacokinetic Parameter: Cmax/D
Description: Maximum observed plasma concentration divide by topical dose (Cmax/D) of paromomycin following administration of paromomycin alone or WR 279,396 to adults in Panama
Time Frame: 0, 0.5, 1.0, 2.0, 3.0, 4.0, 8.0, 12.0, 24.0 hours on both Days 1 and 20
Population: Adults (18+ years)
Measure: Mean (Standard Deviation); unit: 1/ML
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Number analyzed (Participants) | 5 | 4
1/ML
  Day 1 | 185 (144) | 45.9 (35.8)
  Day 20 | 368 (196) | 283 (118)

9. Secondary Outcome: Pharmacokinetic Parameter: AUC/D
Description: Area under the plasma concentration-time curve over 24 hrs divided by topical dose (AUC/D) of paromomycin following administration of paromomycin alone or WR 279,396 to adults in Panama
Time Frame: Days 1 and 20
Population: Adults (18+ years)
Measure: Mean (Standard Deviation); unit: hr/ML
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Number analyzed (Participants) | 5 | 4
hr/ML
  Day 1 | 996.7 (976.1) | 340.5 (368.9)
  Day 20 | 3335 (1482) | 3155 (2151)

10. Secondary Outcome: Final Clinical Cure on All Lesions Independent of Subjects
Description: Final clinical cure was defined as follows:
  1. Subject has initial clinical cure (100% re-epithelialization of lesion by nominal Day 63); OR,
  2. Subject has initial clinical improvement (> 50% re-epithelialization of lesion by nominal Day 63 followed by 100% re-epithelialization of the lesion on or before nominal Day 100; AND,
  3. Subject has no relapse of lesion by Day 168. Relapse was defined as a lesion meeting the criteria for initial clinical cure that had any new ulceration/nodule (> 0 x 0 mm measurement) by nominal day 168, or a lesion meeting the criteria for initial clinical improvement that subsequently enlarged by nominal Day 168.
Time Frame: Initial clinical cure by day 63 and no relapse by day 168
Measure: Number; unit: Cured ulcerated lesions
Units Other Than Participants: Total number of ulerated lesions
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Number analyzed (Participants) | 16 | 14
Number analyzed (Total number of ulerated lesions) | 22 | 21
Cured ulcerated lesions | 12 | 14

11. Secondary Outcome: Number of Index Lesions Meeting Criteria for Clinical Cure During the Study
Description: Number of study participants who meet the criteria for clinical cure (100% re-epithelialization) at specified timepoints during the study.
Time Frame: Day 1, 4, 7, 12, 17, 20, 28, 35, 42, 49, 56, 63, 100, 168
Measure: Number; unit: Lesions meeting clinical cure criteria
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Number analyzed (Participants) | 16 | 14
Lesions meeting clinical cure criteria
  Day 1 | 0 | 0
  Day 4 | 0 | 0
  Day 7 | 0 | 0
  Day 12 | 0 | 0
  Day 17 | 0 | 0
  Day 20 | 1 | 0
  Day 28 | 5 | 6
  Day 35 | 8 | 11
  Day 42 | 10 | 11
  Day 49 | 10 | 12
  Day 56 | 11 | 10
  Day 63 | 11 | 10
  Day 100 | 12 | 10
  Day 168 | 11 | 9

ADVERSE EVENTS:
Arm/Group | Paromomycin Alone Treatment | WR 279,396
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 16/16 | 14/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paromomycin Alone Treatment (N=16) | WR 279,396 (N=14)
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 2
Motion sickness (Ear and labyrinth disorders) | 0 | 1
Bleeding anovulatory (Endocrine disorders) | 0 | 1
Conjunctivitis allergic (Eye disorders) | 1 | 1
Myopia (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Lip dry (Gastrointestinal disorders) | 0 | 1
Application site bleeding (General disorders) | 2 | 2
Application site erythema (General disorders) | 12 | 9
Application site induration (General disorders) | 2 | 1
Application site oedema (General disorders) | 6 | 5
Application site pain (General disorders) | 13 | 3
Application site papules (General disorders) | 1 | 1
Application site pruritus (General disorders) | 16 | 14
Application site vesicles (General disorders) | 2 | 6
Injection site extravasation (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 12 | 11
Application site cellulitis (Infections and infestations) | 0 | 1
Cutaneous leishmaniasis relapse (Infections and infestations) | 2 | 3
Gastroenteritis (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 3
Nasopharyngitis (Infections and infestations) | 1 | 4
Oral herpes (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Superinfection bacterial (Infections and infestations) | 3 | 2
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 12 | 9
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Skin injury (Injury, poisoning and procedural complications) | 1 | 1
Blood triglycerides increased (Investigations) | 0 | 1
Headache (Investigations) | 6 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Burning sensation (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 2
Lymphoedema (Vascular disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Vessel puncture site pain (General disorders) | 1 | 0
Cutaneous leishmaniasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
All randomized subjects were included in the mITT analysis. All subjects also met the criteria for the evaluable subset; therefore, no separate analysis of an evaluable subset of subjects was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Parties agree to keep Referenced Information in strict confidence and not to disclose it to any other party or use Referenced Information for any purpose, other than for the performance of the clinical studies herein described, without prior written consent of the providing party. Parties may disclose the Referenced Information to their employees and consultants, and employees and consultants of their affiliates, who have a need to know such Referenced Information.